CLINICAL TRIAL: NCT06608329
Title: A Randomized, Open-label, Crossover Study to Evaluate Relative Bioavailability, and Food Effect of HDM1002 in Healthy Subjects
Brief Title: A Relative Bioavailability and Food Effect Study of HDM1002 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-108
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy Adult Subject
Keywords: HDM1002 tablet; Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Period 1: Subjects received HDM1002 table (200 mg×1）in fasted state; Period 2: Subjects received HDM1002 tables (100 mg×2）in fasted state; Period 3: Subjects received HDM1002 table (200 mg×1）in fed state.
  Interventions: Drug: HDM1002
- Cohort 2 (Experimental): Period 1: Subjects received HDM1002 tables (100 mg×2）in fasted state; Period 2: Subjects received HDM1002 table (200 mg×1）in fed state; Period 3: Subjects received HDM1002 table (200 mg×1）in fasted state.
  Interventions: Drug: HDM1002
- Cohort 3 (Experimental): Period 1: Subjects received HDM1002 table (200 mg×1）in fed state; Period 2: Subjects received HDM1002 table (200 mg×1）in fasted state; Period 3: Subjects received HDM1002 tables (100 mg×2）in fasted state.
  Interventions: Drug: HDM1002

INTERVENTIONS:
Drug: HDM1002 — Single dose, administered orally. The study is a randomized, open-label, single dose, 3-period, 3 sequence, crossover design.

SUMMARY:
The main purpose of this study is to evaluate the effect of formulation on relative bioavailability of HDM1002, and the food effect on pharmacokinetics of HDM1002.

ELIGIBILITY:
Inclusion Criteria:

1. According to the medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination results during the screening period, the investigator considers the subject to be in good general health.
2. Age range of 18-45 years old (including range), no limit to gender.
3. Male subject weighed ≥50.0 kg, female subject weighed ≥45.0 kg, and a body mass index (BMI) within the range of 19.0 - 30.0 kg/m2 (including cut-off values).
4. Female subject of childbearing potentiaafter last dose, who have no childbearing plans and agrl during signature ICF to 30 days after last dose and male subject during signature ICF to 90 days ee to use highly effective contraception and consent not to donate sperm and oocyte during this period.

Exclusion Criteria:

1. Subject has a history or family history of medullary thyroid cancer, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2), or calcitonin≥50 ng/L during the screening period.
2. History of chronic pancreatitis or an episode of acute pancreatitis within 3 months prior to screening.
3. History of acute cholecystitis attack within 3 months prior to screening.
4. Subject judged by investigator has dysphagia, diseases or conditions that affect gastric emptying, or affect the absorption of gastrointestinal nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, etc.
5. History of previous surgery that will affect the absorption, distribution, metabolism, and excretion of drugs or plan to undergo surgery during the study period.
6. During screening period, any abnormalities in physical examination, electrocardiogram, laboratory tests, and vital signs which are of clinically significant .
7. Taken or planned to take any drug that effect liver enzyme or transporter activity within 28 days prior to taking the investigational drug.
8. History of clinically significant cardiovascular and cerebrovascular disease within 6 months prior to screening or at the time of admission.
9. Presence of clinically significant ECG results judged by the investigator at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
AUC[0-∞] | Day1-Day17
  Area under the curve from time 0 hour to ∞
AUC[0-t] | Day1-Day17
  Area under the curve from time 0 to t hour
Cmax | Day1-Day17
  Maximum observed concentration
Tmax | Day1-Day17
  Time to maximum plasma concentration
t1/2 | Day1-Day17
  Half life
CL/F | Day1-Day17
  Apparent Clearance
Vz/F | Day1-Day17
  Apparent volume of distribution
F | Day1-Day17
  Relative Bioavailability

SECONDARY OUTCOMES:
Adverse events (AEs) | Day1-Day17
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China